CLINICAL TRIAL: NCT01961414
Title: Treat and Extend Therapy Using Intravitreal Aflibercept (IAI) for Previously Treated Patients Exiting the Wet Age-related Macular Degeneration Extension Study (0910)
Brief Title: Treat and Extend Therapy Study Using Intravitreal Aflibercept for Patients Exited From Protocol VGFT-OD 0910
Acronym: RANGE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Palmetto Retina Center, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFT-OD-1319
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: Exudative; AMD; Macular; Degeneration; Aflibercept; Eylea; Intravitreal
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (Experimental): All patients will receive aflibercept 2.0mg intravitreal injection
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Patients will receive Aflibercept 2.0mg intravitreal injection at all scheduled study visits
  Other Names: Eylea 2.0mg, VEGF TRAP-EYE

SUMMARY:
The purpose of this research study is to determine if a "Treat and Extend" regimen (increasing the time between visits when the disease is stable and not getting worse) of aflibercept 2.0mg injections inside the eye for treating patients with Wet Age-related Macular Degeneration.

DETAILED DESCRIPTION:
After exiting VGFT-OD 0910, patients will be enrolled into RANGE, a longterm extension trial evaluating the safety and efficacy of aflibercept IAI utilizing a "treat and extend" regimen. Using pre-specified re-treatment criteria, treatment intervals will be variable with dosing of the active treatment at least every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Previous enrollment in 0910-extension study evaluating intravitreal aflibercept injection (NCT 00964795) without early study discontinuation prior to sponsor early termination.
* Patients are enrolled within 90 days of site activation (all attempts will be made to ensure IAI is given once exited from the 0910-extension and prior to enrollment).
* Willing and able to comply with clinical visits and study related procedures.
* Provide signed informed consent

Exclusion Criteria:

* Prior treatment with verteporfin, or external-beam radiation therapy, or transpupillary thermotherapy in the study eye
* Previous subfoveal focal laser photocoagulation involving the foveal center in the study eye
* History of vitrectomy, submacular surgery, or other surgical intervention for AMD in the study eye
* Any concurrent intraocular condition in the study eye (e.g. diabetic retinopathy or glaucoma) that, in the opinion of the investigator, could either

  * require medical or surgical intervention during the study period to prevent or treat visual loss that might result from that condition, or
  * if allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of best corrected visual acuity over the study period
* Active intraocular inflammation (grade trace or above) in the study eye, or history of idiopathic or autoimmune-associated uveitis in either eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia, ACIOL, or unstable PCIOL
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥30 mmHg despite treatment with anti-glaucoma medication)
* Pregnant or breast-feeding women
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)

  * Contraception is not required for men with documented vasectomy.

    * Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Portion of patients who maintain vision (loss of < or = 5 letters ETDRS BCVA) from baseline to Year 1. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: William L. Clark, M.D., Principal Investigator — Palmetto Retina Center, LLC
Locations (6):
- United States (6):
  - Southeast Retina, Augusta, Georgia
  - Eye Surgical Associates, Lincoln, Nebraska
  - Palmetto Retina Center, West Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Retina Consultants Houston, Houston, Texas
  - Rocky Mountain Retina, Salt Lake City, Utah